CLINICAL TRIAL: NCT00331851
Title: Liraglutide Effect and Action in Diabetes (LEAD-5): Effect on Glycaemic Control After Once Daily Administration of Liraglutide in Combination With Glimepiride and Metformin Versus Glimepiride and Metformin Combination Therapy, and Versus Insulin Glargine Added to Glimepiride and Metformin Combination Therapy in Subjects With Type 2 Diabetes.A Six-month Randomised, Double-blind, Parallel-group, Multi-centre, Multi-national Trial With an Open-label Treat-to-target Insulin Glargine Control Arm.
Brief Title: Effect of Liraglutide on Blood Glucose Control in Subjects With Type 2 Diabetes
Acronym: LEAD-5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1697
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; Insulin Glargine; Metformin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: liraglutide
Drug: insulin glargine
Drug: metformin
Drug: glimepiride

SUMMARY:
This trial is conducted in Africa, Asia, Europe and South America. This trial is designed to show the effect of treatment with liraglutide added to existing glimepiride and metformin combination therapy and to compare it with the effects of insulin glargine added to combination therapy of glimepiride and metformin.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Treatment with oral anti-diabetic drugs for at least 3 months
* HbA1c: 7.5-10.0 % (both incl.) in subjects on OAD monotherapy. 7.0-10.0 % (both incl.) in subjects on OAD combination therapy.
* Body Mass Index (BMI) less than or equal to 45 kg/m2

Exclusion Criteria:

* Treatment with insulin within the last 3 months
* Treatment with any drug that could interfere with the glucose level
* Any serious medical condition
* Females who are pregnant, have intention of becoming pregnant or are breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Actual)
Dates: Start 2006-05; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 26 weeks of treatment

SECONDARY OUTCOMES:
body weight
Safety and tolerability
Beta-cell function
Glycaemic control

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (102):
- Argentina (5):
  - Novo Nordisk Investigational Site, Bahía Blanca
  - Novo Nordisk Investigational Site, Ciudad Autonoma de Bs As
  - Novo Nordisk Investigational Site, Junín
  - Novo Nordisk Investigational Site, Mendoza
  - Novo Nordisk Investigational Site, Rosario
- Austria (2):
  - Novo Nordisk Investigational Site, Bregenz
  - Novo Nordisk Investigational Site, Vienna
- Brazil (3):
  - Novo Nordisk Investigational Site, Curitiba
  - Novo Nordisk Investigational Site, Rio de Janeiro
  - Novo Nordisk Investigational Site, São Paulo
- Denmark (7):
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, Esbjerg
  - Novo Nordisk Investigational Site, Gentofte Municipality
  - Novo Nordisk Investigational Site, Hellerup
  - Novo Nordisk Investigational Site, Hillerød
  - Novo Nordisk Investigational Site, Roskilde
  - Novo Nordisk Investigational Site, Slagelse
- Finland (4):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Kuopio
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, Turku
- France (9):
  - Novo Nordisk Investigational Site, Besançon
  - Novo Nordisk Investigational Site, Brest
  - Novo Nordisk Investigational Site, Corbeil-Essonnes
  - Novo Nordisk Investigational Site, Dijon
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Nanterre
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Nevers
  - Novo Nordisk Investigational Site, Vénissieux
- India (5):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Karnāl, Haryana
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, Hyderabad
  - Novo Nordisk Investigational Site, Patna
- Italy (10):
  - Novo Nordisk Investigational Site, Bergamo
  - Novo Nordisk Investigational Site, Bologna
  - Novo Nordisk Investigational Site, Catania
  - Novo Nordisk Investigational Site, Catanzaro
  - Novo Nordisk Investigational Site, Chieri
  - Novo Nordisk Investigational Site, Chieti Scalo
  - Novo Nordisk Investigational Site, Messina
  - Novo Nordisk Investigational Site, Padua
  - Novo Nordisk Investigational Site, Parma
  - Novo Nordisk Investigational Site, Siena
- Netherlands (8):
  - Novo Nordisk Investigational Site, Almere Stad
  - Novo Nordisk Investigational Site, Den Helder
  - Novo Nordisk Investigational Site, Eindhoven
  - Novo Nordisk Investigational Site, Gouda
  - Novo Nordisk Investigational Site, Maastricht
  - Novo Nordisk Investigational Site, The Hague
  - Novo Nordisk Investigational Site, Zevenaar
  - Novo Nordisk Investigational Site, Zoetermeer
- Norway (7):
  - Novo Nordisk Investigational Site, Bergen
  - Novo Nordisk Investigational Site, Gjettum
  - Novo Nordisk Investigational Site, Jessheim
  - Novo Nordisk Investigational Site, Nordbyhagen
  - Novo Nordisk Investigational Site, Notodden
  - Novo Nordisk Investigational Site, Sandvika
  - Novo Nordisk Investigational Site, Skedsmokorset
- Philippines (4):
  - Novo Nordisk Investigational Site, Cebu City
  - Novo Nordisk Investigational Site, Manila
  - Novo Nordisk Investigational Site, Marikina City
  - Novo Nordisk Investigational Site, Pasig
- Poland (6):
  - Novo Nordisk Investigational Site, Gdynia
  - Novo Nordisk Investigational Site, Katowice
  - Novo Nordisk Investigational Site, Opole
  - Novo Nordisk Investigational Site, Poznan
  - Novo Nordisk Investigational Site, Wroclaw
  - Novo Nordisk Investigational Site, Zabrze
- Novo Nordisk Investigational Site, Moscow, Russia
- Serbia and Montenegro (2):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Nis
- Slovakia (6):
  - Novo Nordisk Investigational Site, Banská Bystrica
  - Novo Nordisk Investigational Site, Bratislava
  - Novo Nordisk Investigational Site, L'ubochna
  - Novo Nordisk Investigational Site, Martin
  - Novo Nordisk Investigational Site, Nitra
  - Novo Nordisk Investigational Site, Žilina
- South Africa (3):
  - Novo Nordisk Investigational Site, Bloemfontein, Free State
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Worcester, Western Cape
- Spain (8):
  - Novo Nordisk Investigational Site, Barakaldo
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Getafe
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Santiago de Compostela
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valencia
  - Novo Nordisk Investigational Site, Valladolid
- United Kingdom (12):
  - Novo Nordisk Investigational Site, Ayr
  - Novo Nordisk Investigational Site, Bradford
  - Novo Nordisk Investigational Site, Guildford
  - Novo Nordisk Investigational Site, Liverpool
  - Novo Nordisk Investigational Site, Livingstone
  - Novo Nordisk Investigational Site, Llantrisant
  - Novo Nordisk Investigational Site, Manchester
  - Novo Nordisk Investigational Site, Nottingham
  - Novo Nordisk Investigational Site, Salford
  - Novo Nordisk Investigational Site, Sheffield
  - Novo Nordisk Investigational Site, Swansea
  - Novo Nordisk Investigational Site, Watford

REFERENCES:
- [Result] Sullivan SD, Alfonso-Cristancho R, Conner C, Hammer M, Blonde L. Long-term outcomes in patients with type 2 diabetes receiving glimepiride combined with liraglutide or rosiglitazone. Cardiovasc Diabetol. 2009 Feb 26;8:12. doi: 10.1186/1475-2840-8-12. PMID 19245711
- [Result] McGill JB. Insights from the Liraglutide Clinical Development Program--the Liraglutide Effect and Action in Diabetes (LEAD) studies. Postgrad Med. 2009 May;121(3):16-25. doi: 10.3810/pgm.2009.05.1998. PMID 19491536
- [Result] Russell-Jones D, Vaag A, Schmitz O, Sethi BK, Lalic N, Antic S, Zdravkovic M, Ravn GM, Simo R; Liraglutide Effect and Action in Diabetes 5 (LEAD-5) met+SU Study Group. Liraglutide vs insulin glargine and placebo in combination with metformin and sulfonylurea therapy in type 2 diabetes mellitus (LEAD-5 met+SU): a randomised controlled trial. Diabetologia. 2009 Oct;52(10):2046-55. doi: 10.1007/s00125-009-1472-y. Epub 2009 Aug 14. PMID 19688338
- [Result] Blonde L, Russell-Jones D. The safety and efficacy of liraglutide with or without oral antidiabetic drug therapy in type 2 diabetes: an overview of the LEAD 1-5 studies. Diabetes Obes Metab. 2009 Dec;11 Suppl 3:26-34. doi: 10.1111/j.1463-1326.2009.01075.x. PMID 19878259
- [Result] Buse JB, Garber A, Rosenstock J, Schmidt WE, Brett JH, Videbaek N, Holst J, Nauck M. Liraglutide treatment is associated with a low frequency and magnitude of antibody formation with no apparent impact on glycemic response or increased frequency of adverse events: results from the Liraglutide Effect and Action in Diabetes (LEAD) trials. J Clin Endocrinol Metab. 2011 Jun;96(6):1695-702. doi: 10.1210/jc.2010-2822. Epub 2011 Mar 30. PMID 21450987
- [Result] Bode BW, Brett J, Falahati A, Pratley RE. Comparison of the efficacy and tolerability profile of liraglutide, a once-daily human GLP-1 analog, in patients with type 2 diabetes >/=65 and <65 years of age: a pooled analysis from phase III studies. Am J Geriatr Pharmacother. 2011 Dec;9(6):423-33. doi: 10.1016/j.amjopharm.2011.09.007. Epub 2011 Nov 4. PMID 22055210
- [Result] Henry RR, Buse JB, Sesti G, Davies MJ, Jensen KH, Brett J, Pratley RE. Efficacy of antihyperglycemic therapies and the influence of baseline hemoglobin A(1C): a meta-analysis of the liraglutide development program. Endocr Pract. 2011 Nov-Dec;17(6):906-13. doi: 10.4158/ep.17.6.906. PMID 22193143
- [Result] Zinman B, Schmidt WE, Moses A, Lund N, Gough S. Achieving a clinically relevant composite outcome of an HbA1c of <7% without weight gain or hypoglycaemia in type 2 diabetes: a meta-analysis of the liraglutide clinical trial programme. Diabetes Obes Metab. 2012 Jan;14(1):77-82. doi: 10.1111/j.1463-1326.2011.01493.x. Epub 2011 Oct 30. PMID 21883806
- [Result] Niswender K, Pi-Sunyer X, Buse J, Jensen KH, Toft AD, Russell-Jones D, Zinman B. Weight change with liraglutide and comparator therapies: an analysis of seven phase 3 trials from the liraglutide diabetes development programme. Diabetes Obes Metab. 2013 Jan;15(1):42-54. doi: 10.1111/j.1463-1326.2012.01673.x. Epub 2012 Sep 9. PMID 22862847
- [Result] Alves C, Batel-Marques F, Macedo AF. A meta-analysis of serious adverse events reported with exenatide and liraglutide: acute pancreatitis and cancer. Diabetes Res Clin Pract. 2012 Nov;98(2):271-84. doi: 10.1016/j.diabres.2012.09.008. Epub 2012 Sep 23. PMID 23010561
- [Result] King AB, Montanya E, Pratley RE, Blonde L, Svendsen CB, Donsmark M, Sesti G. Liraglutide achieves A1C targets more often than sitagliptin or exenatide when added to metformin in patients with type 2 diabetes and a baseline A1C <8.0%. Endocr Pract. 2013 Jan-Feb;19(1):64-72. doi: 10.4158/EP12232.OR. PMID 23186975
- [Result] Buse JB, Peters A, Russell-Jones D, Furber S, Donsmark M, Han J, MacConell L, Maggs D, Diamant M. Is insulin the most effective injectable antihyperglycaemic therapy? Diabetes Obes Metab. 2015 Feb;17(2):145-51. doi: 10.1111/dom.12402. Epub 2014 Nov 9. PMID 25323312
- [Result] Jensen TM, Saha K, Steinberg WM. Is there a link between liraglutide and pancreatitis? A post hoc review of pooled and patient-level data from completed liraglutide type 2 diabetes clinical trials. Diabetes Care. 2015 Jun;38(6):1058-66. doi: 10.2337/dc13-1210. Epub 2014 Dec 12. PMID 25504028
- [Derived] Fonseca VA, Devries JH, Henry RR, Donsmark M, Thomsen HF, Plutzky J. Reductions in systolic blood pressure with liraglutide in patients with type 2 diabetes: insights from a patient-level pooled analysis of six randomized clinical trials. J Diabetes Complications. 2014 May-Jun;28(3):399-405. doi: 10.1016/j.jdiacomp.2014.01.009. Epub 2014 Jan 21. PMID 24561125
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com